CLINICAL TRIAL: NCT04140487
Title: A Phase I/II Study of Azacitidine, Venetoclax, and Gilteritinib for Patients With Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome With an Activating FLT3 Mutation
Brief Title: Azacitidine, Venetoclax, and Gilteritinib in Treating Patients With Recurrent/Refractory FLT3-Mutated Acute Myeloid Leukemia, Chronic Myelomonocytic Leukemia, or High-Risk Myelodysplastic Syndrome/Myeloproliferative Neoplasm
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0366; NCI-2019-04959 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0366 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-08-19; First posted 2019-10-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Myelodysplastic/Myeloproliferative Neoplasm; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelomonocytic Leukemia; Refractory Myelodysplastic/Myeloproliferative Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic-Myeloproliferative Diseases | interventions — Azacitidine; gilteritinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (azacitidine, venetoclax, gilteritinib) (Experimental): Patients receive azacitidine SC or IV over 30-60 minutes on days 1-7, venetoclax PO QD on days 1-28 of cycle 1 and on days 1-21 of subsequent cycles, and gilteritinib PO QD on days 1-28. Treatment of azacytidine and venetoclax repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Cycles of gilteritinib repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Azacitidine; Drug: Gilteritinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; Onureg; U-18496; Vidaza
Drug: Gilteritinib — Given PO
  Other Names: ASP-2215; ASP2215
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I/II trial studies the side effects and best dose of gilteritinib and to see how well it works in combination with azacitidine and venetoclax in treating patients with FLT3-mutation positive acute myeloid leukemia, chronic myelomonocytic leukemia, or high-risk myelodysplastic syndrome/myeloproliferative neoplasm that has come back (recurrent) or has not responded to treatment (refractory). Drugs used in chemotherapy, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Venetoclax may stop the growth of cancer cells by blocking Bcl-2, a protein needed for cancer cell survival. Gilteritinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving azacitidine, venetoclax, and gilteritinib may work better compared to azacitidine and venetoclax alone in treating patients with acute myeloid leukemia, chronic myelomonocytic leukemia, or myelodysplastic syndrome/myeloproliferative neoplasm.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) of the combination of azacitidine, venetoclax and gilteritinib in patients with relapsed/refractory FLT3-mutated acute myeloid leukemia (AML) or chronic myelomonocytic leukemia (CMML) or high-risk myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN). (Phase I) II. To determine the complete remission/complete remission with incomplete count recovery (CR/CRi) rate of the regimen in patients with newly diagnosed or relapsed/refractory fms-like tyrosine kinase 3 (FLT3)-mutated AML or CMML or high-risk MDS/MPN. (Phase II)

SECONDARY OBJECTIVES:

I. To assess other efficacy endpoints (CR rate, minimal residual disease negativity by flow cytometry, relapse-free survival, overall survival).

II. To assess proportion of patients proceeding to hematopoietic stem cell transplantation (HSCT).

III. To determine the safety of the combination regimen.

EXPLORATORY OBJECTIVES:

I. To evaluate the impact of baseline genomic alterations on response and survival of the combination regimen.

II. To determine the impact of baseline FLT3 allelic ratio on response and survival.

III. To evaluate clonal evolution from diagnosis to relapse using single-cell sequencing.

OUTLINE: This is phase I, dose-escalation study of gilteritinib followed by a phase II study.

Patients receive azacitidine subcutaneously (SC) or intravenously (IV) over 30-60 minutes on days 1-7, venetoclax orally (PO) once daily (QD) on days 1-28 of cycle 1 and on days 1-21 of subsequent cycles, and gilteritinib PO QD on days 1-28. Treatment of azacytidine and venetoclax repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Cycles of gilteritinib repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

  * Phase I cohort: Adults ≥ 18 years with relapsed/refractory FLT3-mutated AML or CMML or other MDS/MPN that is intermediate-2 or high-risk by the International Prognostic Scoring System
  * Phase II cohort A: Adults ≥ 18 years with newly diagnosed FLT3-mutated AML
  * Phase II cohort B: Adults ≥ 18 years with relapsed/refractory FLT3-mutated AML or CMML or other MDS/MPN that is intermediate-2 or high-risk by the International Prognostic Scoring System
  * For all cohorts, patients with either FLT3-internal tandem duplication (FLT3-ITD) or FLT3 D835 mutations will be eligible
* Performance status ≤ 3 (Eastern Cooperative Oncology Group [ECOG] scale)
* Total serum bilirubin ≤ 2.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, hemolysis or the underlying leukemia approved by the principal investigator (PI)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 3 x ULN, unless due to the underlying leukemia approved by the PI
* Creatinine clearance ≥ 30 mL/min
* Ability to swallow
* Signed informed consent

Exclusion Criteria:

* Prior therapies:

  * Phase I cohort: No restriction based on prior therapies
  * Phase II cohort A: Patients with prior therapy for AML are not eligible. Prior therapy for antecedent hematologic disorder is allowed. Prior hydroxyurea or cytarabine given for purposes of cytoreduction is also allowed. Prior all trans-retinoic acid given for presumed acute promyelocytic leukemia is also allowed
  * Phase II cohort B: No restriction on number of prior therapies
* Patients suitable for and willing to receive intensive induction chemotherapy (for Phase II cohort A only)
* Congenital long QT syndrome or corrected QT interval by Fridericia (QTcF) > 450 msec. Repeat electrocardiograms (EKGs) after correction of electrolytes or discontinuation of QT prolonging medications are allowed to meet entry criteria. In cases where QTcF > 450 msec is considered to be falsely increased due to inaccurate automated reading and not clinically significant (e.g. due to bundle branch block), patients are still eligible if cardiologist reviews and documents that QTcF is ≤ 450 msec when manually measured
* Active serious infection not controlled by oral or intravenous antibiotics (e.g. persistent fever or lack of improvement despite antimicrobial treatment)
* Active grade III-V cardiac failure as defined by the New York Heart Association criteria
* Active central nervous system leukemia
* Known human immunodeficiency virus (HIV) seropositive
* Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection

  * Note: Patients who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment is not anticipated to interfere with the safety or efficacy assessment of the investigational regimen may be included only after discussion with the PI
* Consumed strong inducer of cytochrome P450, family 3, subfamily A (CYP3A) or p-glycoprotein within 3 days of study enrollment. Agents include but are not limited to: carbamazepine, phenytoin, rifampin, and St. John's wort
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Prior recent treatment with corticosteroids, hydroxyurea and/or cytarabine (given for cytoreduction) permitted
* Pregnant women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception throughout the study period and for at least 6 months after the last dose of study drugs. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control throughout the study period and for at least 4 months after the last dose of study drugs. Lactating women (or those planning to breastfeed) should not breastfeed during treatment of gilteritinib and for at least 2 months after the last dose of gilteritinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of gilteritinib (Phase I) | Up to 28 days
  The MTD is the highest dose level in which < 2 patients of 6 develop first cycle dose-limiting toxicity.
Overall response rate (OR) (Phase II) | Up to 56 days (2 cycles)
  Will be defined as the complete remission/complete remission with incomplete count recovery (CR/CRi) rate. Will estimate the OR for the combination treatment along with the 95% credible interval.

SECONDARY OUTCOMES:
Complete response rate | Up to 3 years
  Will be estimated along with 95% credible interval.
Minimal residual disease negativity | Up to 3 years
  Will be assessed by flow cytometry and estimated along with 95% credible interval.
Relapse-free survival | The number of days from the date of response to the date of documented relapses from CR or death from any cause, whichever occurs first, assessed up to 3 years
  Will be estimated using the method of Kaplan and Meier.
Overall survival | From the start of treatment until death or last follow-up, assessed for up to 3 years
  Will be estimated using the method of Kaplan and Meier.
Proportion of patients proceeding to hematopoietic stem cell transplantation | Up to 3 years
  Will be estimated along with 95% credible interval.
Incidence of adverse events | Up to 3 years
  Will be summarized using descriptive statistics such as mean, standard deviation, median and range.

OTHER OUTCOMES:
Impact of genomic alterations | Baseline
  The impact of genomic alterations on response and the survival of the combination regimen will be assessed. Will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Impact of FLT3 allelic ratio | Baseline
  The impact of FLT3 allelic ratio on response and the survival will be assessed. Will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Minimal residual disease negativity rates | At time of remission
  Will be assessed by digital droplet polymerase chain reaction. Will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.
Evaluation of leukemia stem cell populations | Up to 3 years
  Will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Short NJ, Daver N, Dinardo CD, Kadia T, Nasr LF, Macaron W, Yilmaz M, Borthakur G, Montalban-Bravo G, Garcia-Manero G, Issa GC, Chien KS, Jabbour E, Nasnas C, Huang X, Qiao W, Matthews J, Stojanik CJ, Patel KP, Abramova R, Thankachan J, Konopleva M, Kantarjian H, Ravandi F. Azacitidine, Venetoclax, and Gilteritinib in Newly Diagnosed and Relapsed or Refractory FLT3-Mutated AML. J Clin Oncol. 2024 May 1;42(13):1499-1508. doi: 10.1200/JCO.23.01911. Epub 2024 Jan 26. PMID 38277619
- See also: Related Info — http://www.mdanderson.org